CLINICAL TRIAL: NCT04137146
Title: Sacral Nerve Stimulation in the Treatment of Gait Disorder in Patients With Parkinson's Disease
Brief Title: SNS for Treatment of PD Gait Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bomin Sun, Bomin Sun, Chief physician, Ruijin Hospital, Ruijin Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2019 SNS for gait disturbance
Record Dates: First submitted 2019-10-18; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacral Nerve Stimulation (Experimental): Intervention: Sacral nerve Stimulation Stimulation sites：S3 Postoperative study visits lasted approximately 3 hours and were conducted in 3 months.
  Interventions: Device: Sacral Nerve Stimulation
- No SNS Intervention (No Intervention)

INTERVENTIONS:
Device: Sacral Nerve Stimulation — Implantation of a sacral nerve neurostimulation system: A single electrode (Interstim® model 3889-28; Medtronic, Minneapolis, MN) was inserted bilaterally into the sacral foramen (S3), connected to an internal pulse generator (Medtronic Interstim
  ® II 3058)
  Arms: Sacral Nerve Stimulation

SUMMARY:
Parkinson's disease (PD) is a progressive disease, characterized by dopaminergic neurons degeneration in the substantia nigra. Postural and gait disorders usually occur in advanced PD patients. However, existing drugs and deep brain stimulation (DBS) therapy are not effective enough for these axial symptoms or cannot maintain long-term efficacy, which seriously reduce patients' quality of life. Sacral nerve stimulation(SNS) is a treatment for urinary symptoms in PD. It has been reported that SNS can also improve PD gait disturbance, but the level of evidence currently is low. We assume that SNS may have a similar mechanism to spinal cord stimulation and may be an effective treatment for PD gait disorder. However, there are few studies on the mechanism of SNS treatment. Therefore, we will conduct a large sample, prospective case-control study to provide a higher level of clinical evidence for sacral nerve stimulation in the treatment of gait disturbance in PD. Our primary objective is to evaluate the efficacy of SNS for gait disorder in PD. PD patients who have received DBS surgery but still have severe gait problems will be included. This study will contribute to evaluate the efficacy of SNS for gait disorder in PD, provide level II evidence for expanding the indications of SNS, varicocelectomy., and improve patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease, Hoehn & Yahr stage (medication off condition) at 2~4;
* Gait and balance disorder, unstable posture, frequently falls (gaze and fall questionnaire (GFQ) score > 32) and severe dysuria, extremely affects quality of life (overactive bladder score (OABSS) ≥12);
* SCS eligibility has been confirmed by neurologist and neurosurgeon;
* Patients willingly seek surgical treatment for PD gait disturbance；
* Ability to perform a gait/walking task (under close supervision);
* Informed consent and have good compliance.

Exclusion Criteria:

* Lesion in spinal nerve or other surgical contraindications;
* Severe depression (Beck Depression Inventory scores > 25) or dementia (Mini Mental State Examination < 24);
* Medical history of stroke, amyotrophic lateral sclerosis or myasthenia gravis;
* Other neuropsychiatric disorders or relevant medical history;
* Taking prohibited medications (such as lithium, valproate, steroids, adrenergic agonists, etc.);
* Cardiac, renal or other important organs hypofunction or dysfunction, or unstable vital signs;
* Women reporting that they are pregnant;
* Any situation (medical, psychological, social, geographical, etc.) that may endanger patient's life or result in patients withdrawing from the study at present or in the future.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Parameter changes in Timed Up and Go Test | Baseline (preoperative), during external test stimulation (1-14 days after electrode implantation), 3 months post-SNS
  Patients should stand up from the chair, walk forward for 3m with daily speed, turn after passing the marked line, and then walk back to the chair and sit down, leaning back in the chair. Video recordings will be made throughout the test.

SECONDARY OUTCOMES:
Changes in Uniﬁed Parkinson's Disease Rating Scale Part Ⅲ (UPDRS Ⅲ) scores | Baseline (preoperative), 3 months post-SNS
  Uniﬁed Parkinson's Disease Rating Scale Part Ⅲ (UPDRS Ⅲ) measures the motor severity of Parkinson's disease. UPDRS Ⅲ score has a range of 0 (no symptoms) to 132 (severe disease symptoms).
Changes in Gait and Fall Questionnaire (GFQ) scores | Baseline (preoperative), 3 months post-SNS
  GFQ is a subjective scale for gait problems in the past 4 weeks. GFQ score has a range of 0 (no gait problems) to 64 (severe gait problems)
Changes in Berg Balance scale (BBS) scores | Baseline (preoperative), 3 months post-SNS
  BBS measures patients' static and dynamic balance abilities. BBS score has a range of 0 (severe balance problems) to 56 (no balance problems).
Changes in 8-item Parkinson's Disease Questionnaire (PDQ-8) scores | Baseline (preoperative), 3 months post-SNS
  PDQ-8 is a reliable and feasible tool for the assessment of quality of life in Parkinson's disease patients.
Changes in EuroQol-5 Dimensions (EQ-5D) scores | Baseline (preoperative), 3 months post-SNS
  EQ-5D measures five dimensions of PD patients' quality of life: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Changes in Montreal cognitive assessment (MoCA) scores | Baseline (preoperative), 3 months post-SNS
  The MoCA is a widely used screening assessment for detecting cognitive impairment. MoCA score has a range of 0 (severe dementia) to 30 (cognitive intact).
Changes in Voiding Diary | Baseline (preoperative), during external test stimulation (1-14 days after electrode implantation), 3 months post-SNS
  The voiding diary recording the patient's daily fluid input and urinary output is a simple but effective tool for assessing storage symptoms.
Parameter changes in Dual task | Baseline (preoperative), 3 months post-SNS
  The protocol requires patient to walk along a walkway of 5 m between two retroreflective markers placed 0.5 m. They are asked to make a left or right turn of 360° around the marker before walking further. They are instruted to complete the task with or without a verbal cognitive color classification task.
Parameter changes in Six-Minute Walking Test | Baseline (preoperative), 3 months post-SNS
  This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes.
Parameter changes in Rapid 360° Turn | Baseline (preoperative), 3 months post-SNS
  The test requires patients to make rapid 360° turns on the spot in both directions.

CONTACTS AND LOCATIONS:
Locations (1):
- Functional neurosurgery of Shanghai jiaotong university affiliated Ruijin hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang C, Wang L, Pan Y, Sun B, Nonnekes J, Bloem BR, Li D. Sacral nerve stimulation improves gait in Parkinson's disease. Brain Stimul. 2019 Jul-Aug;12(4):1075-1076. doi: 10.1016/j.brs.2019.03.074. Epub 2019 Apr 1. No abstract available. PMID 30979641